CLINICAL TRIAL: NCT06818409
Title: Is the CRP-Albumin-Lymphocyte (CALLY) Index Effective in Predicting Postoperative Delirium in Geriatric Patients Undergoing Hip Fracture Surgery
Status: Recruiting | Type: Observational
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, ERBİL TÜRKSAL, Principal Investigator, Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: 2024-BÇEK/195
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Delirium (POD); Hip Fracture; CRP; Albumin; Lymphocyte
MeSH Terms: conditions — Emergence Delirium; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Geriatric patients undergoing hip fracture surgery: Patients aged >65 years undergoing hip fracture surgery during the study period
  Interventions: Diagnostic Test: The Diagnostic and Statistical Manual of Mental Disorders (DSM) - 5 criteria for delirium diagnosis

INTERVENTIONS:
Diagnostic Test: The Diagnostic and Statistical Manual of Mental Disorders (DSM) - 5 criteria for delirium diagnosis — Delirium presence will be assessed using DSM-5 criteria twice daily (morning and evening) for three days, after surgery.

SUMMARY:
Introduction: Postoperative delirium (POD) is a common complication in elderly surgical patients and is significantly associated with prolonged hospital stays, cognitive impairment, functional decline, and increased mortality rates within 6 to 12 months. Its incidence has been reported to range between 10% and 70%, depending on the diagnostic criteria used, the population studied, and the type of surgical procedure performed. The incidence is particularly higher following vascular, cardiac, and hip fracture surgeries.

According to the 2024 updated guidelines by the European Society of Anaesthesiology and Intensive Care (ESAIC), POD should be screened at least once daily for a minimum of three days, beginning in the post-anesthesia recovery unit, based on the DSM-5 criteria. POD is a complex syndrome associated with various phenotypes and is likely the result of a combination of neuroinflammatory and oxidative stress processes.

Candidate biomarkers for POD include inflammatory parameters (such as interleukins, C-reactive protein [CRP], erythrocyte sedimentation rate, and CD68), dopamine receptors, norepinephrine levels, cortisol levels, genetic biomarkers (e.g., apolipoprotein E4), acetylcholinesterase levels, and albumin levels. However, systemic stress can lead to nonspecific activation of the immune system, resulting in a decrease in lymphocyte count.

Although the relationships between CRP, albumin, and lymphocyte count with POD have been individually investigated in the literature, no study has examined the combined effect of these three parameters. Based on this, we aimed to investigate whether the CRP-Albumin-Lymphocyte (CALLY) Index, a novel index not previously reported in the literature, is effective in predicting POD in geriatric patients with hip fractures. The CALLY Index is calculated using the formula: (Albumin × Lymphocyte) / (CRP × 10⁴).

Aim/Hypothesis:

H₀: The CALLY Index cannot predict the risk of postoperative delirium in geriatric patients undergoing hip fracture surgery.

H₁: The CALLY Index can predict the risk of postoperative delirium in geriatric patients undergoing hip fracture surgery.

Material-Methods:

The following data will be recorded for each patient:

* Demographic variables: age, sex, height, weight, and body mass index (BMI)
* American Society of Anesthesiologists (ASA) physical status classification
* Comorbidities and medication use
* Smoking and alcohol consumption history
* Preoperative laboratory parameters: obtained from the hospital information system for CALLY Index calculation
* Perioperative variables: type and duration of anesthesia, duration of surgery, type of surgical procedure, estimated blood loss, blood product transfusion status, and occurrence of intraoperative adverse events
* Postoperative data:
* Ward of admission after surgery (orthopedic ward/intensive care unit)
* Presence of delirium, assessed twice daily (morning and evening) for three days using DSM-5 criteria, starting in the post-anesthesia recovery unit
* Occurrence of postoperative complications
* Length of stay in the intensive care unit
* Total hospital length of stay
* Mortality status

Patients aged 65 years and older who undergo surgery for femoral neck or intertrochanteric fractures will be included in the study. Patients with preoperative delirium, preoperative dementia, pathological or open fractures, systemic or localized infections in the fracture region during the preoperative period, or multiple trauma will be excluded. Additionally, those with a BMI <18.5 or ≥35 chronic organ failure, or advanced-stage cancer will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years and older who undergo surgery for femoral neck or intertrochanteric fractures

Exclusion Criteria:

* Patients with preoperative delirium
* Patients with preoperative dementia
* Patients with pathological fractures
* Patients with open fractures
* Patients with systemic or localized infections in the fracture region during the preoperative period
* Patients with multiple trauma
* Patients with a BMI <18.5 or ≥35
* Patients with chronic organ failure
* Patients with advanced-stage cancer

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: In the literature, the preoperative CRP/albumin ratio has been found to have a sensitivity of 94.1% and a specificity of 43.9% (AUC: 3.69) in detecting postoperative delirium. The incidence of postoperative delirium varies between 10% and 70%, depending on the diagnostic criteria used, the population studied, and the type of surgical procedure. Its incidence is higher following vascular, cardiac, and hip fracture surgeries.
  In our study, which investigates the predictive value of the CRP-Albumin-Lymphocyte (CALLY) Index in detecting delirium after hip fracture in the geriatric patient population, these literature findings were taken into account. Based on the Sample Size Estimation in Diagnostic Accuracy Studies, with a power of 0.85, a Type I error of 5%, a specificity of 43.9%, and a prevalence of 50%, the required sample size was calculated as 84 patients. Considering a 20% margin of error, it was decided to include 100 patients in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2025-08-06 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium | Twice daily (morning and evening) for three days
  Delirium presence will be assessed using DSM-5 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Erbil Türksal, Specialist, Principal Investigator — University of Health Sciences, Ankara Atatürk Sanatorium Training and Research Hospital
Locations (1):
- University of Health Sciences, Ankara Atatürk Sanatorium Training and Research Hospital, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No